CLINICAL TRIAL: NCT04337372
Title: Parent-infant Learning Dynamics During Early Shared Book Reading
Brief Title: Infant and Parent Shared Book Reading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB202000756-N; 1R21HD102715-01 (NIH); 5R21HD102715-02 (NIH)
Record Dates: First submitted 2020-04-02; First posted 2020-04-07 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Individual, Category, and No-label Conditions

STUDY DESIGN:
Intervention Model Description: There were three age groups tested, but all infant-parent dyads were tested on the same conditions and measures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 6 month olds (Active Comparator): 6-month old infants and a parent completed shared book reading and infant visual attention, joint visual attention (dyad, co-occurrence of parent and infant attention toward the book), infant EEG power, and infant-parent EEG coherence were measured in for objects labeled with individual level names, category-level names, and no label. All infant-parent dyads completed all three conditions.
  Interventions: Behavioral: Effects of shared book reading: Labels
- 9 month olds (Active Comparator): 9-month old infants and a parent completed shared book reading and infant visual attention, joint visual attention (dyad, co-occurrence of parent and infant attention toward the book), infant EEG power, and infant-parent EEG coherence were measured in for objects labeled with individual level names, category-level names, and no label. All infant-parent dyads completed all three conditions.
  Interventions: Behavioral: Effects of shared book reading: Labels
- 12 month olds (Active Comparator): 12-month old infants and a parent completed shared book reading and infant visual attention, joint visual attention (dyad, co-occurrence of parent and infant attention toward the book), infant EEG power, and infant-parent EEG coherence were measured in for objects labeled with individual level names, category-level names, and no label. All infant-parent dyads completed all three conditions.
  Interventions: Behavioral: Effects of shared book reading: Labels
- Adult Parents (Active Comparator): Adult parents of infant participants completed shared book reading with their infants. Joint attention and EEG synchrony data were recorded and combined with infant data for analyses. No adult data were analyzed separately from infant data.
  Interventions: Behavioral: Effects of shared book reading: Labels

INTERVENTIONS:
Behavioral: Effects of shared book reading: Labels — Book reading included objects labeled with 1) Individual labels, 2) Category labels, and 3) No Labels. Condition and infant age differences were examined.

SUMMARY:
This work is guided by two specific aims and is expected to result in a better understanding of the effectiveness of shared book reading as a tool for supporting parent-infant interactions and infant learning across the first year of life. This work determined the extent to which books with individually-named characters (e.g., "Boris", "Fiona") increases parent-infant joint attention and infant selective attention relative to books with generic labels (e.g., "Bear", "Bear") or no labels and whether attention differs by age. During infant-parent shared book reading joint attention was measured using dual eye-tracking. Infants and parents then returned to the lab the next day and infant selective attention and infant-parent neural synchrony was measured using EEG.

DETAILED DESCRIPTION:
Shared book reading has been found to have broad developmental benefits for language, socio-emotional and cognitive development. However, the effects of shared book reading on infant development are not well understood. Although healthcare professionals and educators ask parents to read books to their infants early and often, the book reading experience itself has never been systematically investigated in infancy. This work is guided by two specific aims and is expected to result in a better understanding of the effectiveness of shared book reading as a tool for supporting parent-infant interactions and infant learning across the first year of life. The primary aim of the proposed work is to determine the extent to which books with individually-named characters (e.g., "Boris", "Fiona") increases parent-infant joint attention and infant selective attention relative to books with generic labels (e.g., "Bear", "Bear") or no labels and whether attention differs by age. To address the aim of this project, a cross-sectional sample of 6-, 9-, and 12-month old infants and their parents came to the laboratory and read a book that includes three distinct character labeling conditions (individual names, generic category labels, no label). During infant-parent shared book reading joint attention was measured using dual eye-tracking. Infants and parents then returned to the lab the next day and infant selective attention and infant-parent neural synchrony was measured using EEG frequency tagging while infants and their parent viewed familiar characters across labeling conditions as well as unfamiliar characters. This project determined the extent to which parent-infant shared book reading impacted infant attention, parent-infant joint attention, EEG power, and parent-infant EEG synchrony.

ELIGIBILITY:
Inclusion Criteria:

* Infants will be included if they are typically developing and between 5.5 and 12.5 months of age, as well as their caregiver.
* Parents 18-65 years old

Exclusion Criteria:

1. Infants who were born more that 14 days premature.
2. Infants who with a history of neurological or visual deficits.
3. Infants with a history of seizures or a disorder that includes risk of seizures.
4. Infants with a parent that has a history of seizures of a disorder that includes risk of seizures.
5. Parents with a history of seizures or a disorder that includes risk of seizures.

Ages: 5 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Scott, Principal Investigator — University of Florida; Andreas Keil, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Brain, Cognition and Development Laboratory, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and study participation occurred between January 2022 and December 2023 in a research laboratory. Infant participants and their parents came in for two visits within one week, and were not followed up with beyond that.
Groups:
- 6 Month Olds: 6 month olds infants completed the a book reading intervention. A parent and their infant read a short book in the laboratory. Books included three labeling conditions expected to elicit different levels of attention.
- 9 Month Olds: 9 month olds infants completed the a book reading intervention. A parent and their infant read a short book in the laboratory. Books included three labeling conditions expected to elicit different levels of attention.
- 12 Month Olds: 12 month olds infants completed the a book reading intervention. A parent and their infant read a short book in the laboratory. Books included three labeling conditions expected to elicit different levels of attention.
- Adults: Parents of Infants: Data from parents of infants were collected for the joint attention and EEG synchrony task and combined with infant data for analysis. Parent data was not examined separately.
Period: Day 1: Eye-tracking Measures
Arm/Group | 6 Month Olds | 9 Month Olds | 12 Month Olds | Adults: Parents of Infants
Started | 21 (Day 1 included Eye-tracking during shared book reading for infants and parents and infant attention and infant-parent joint attention was measured.) | 26 | 26 | 73
Completed | 20 | 23 | 17 | 60
Not Completed | 1 | 3 | 9 | 13
Not completed — Protocol Violation | 1 | 3 | 7 | 11
Not completed — Equipment Failure | 0 | 0 | 2 | 2
Period: Day 2: EEG Measures
Arm/Group | 6 Month Olds | 9 Month Olds | 12 Month Olds | Adults: Parents of Infants
Started | 21 (Day 2 included EEG data and was analyzed separately from the eye-tracking data. Infants and parents completed an EEG task and infant EEG and infant-parent EEG synchrony were measured.) | 26 | 26 | 73
Completed | 15 | 17 | 19 | 51
Not Completed | 6 | 9 | 7 | 22
Not completed — Lost to Follow-up | 0 | 3 | 2 | 5
Not completed — Protocol Violation | 6 | 6 | 5 | 17

BASELINE CHARACTERISTICS:
Population: 73 infants and their parents (n=146) were recruited. Each dyad (parent-infant) completed shared book reading with books that contain each of the 3 manipulations (individual, category, no label).
Groups:
- Infants: Infants included three groups, 6-month-olds, 9-month-olds, and 12-month-olds.
- Parents: One parent of each infant was included in the dyadic data analysis.
- Total: Total of all reporting groups
Arm/Group | Infants | Parents | Total
Number analyzed (Participants) | 73 | 73 | 146
Age, Categorical [Count of Participants; unit: Participants] — 73 infants and their parents (total n= 146) were recruited and each outcome measure contained different numbers of infants or dyads contributing to the final data set for analysis. 146 is included here as the number of infants and parents recruited. However, 10 infants were lost to follow-up, 2 were tested outside the age window and were then excluded. Additional infants and or parent data was excluded per outcome measure. Population: 73 infants and their parents (n=146) were recruited. Each dyad (parent-infant) completed shared book reading with books that contain each of the 3 manipulations (individual, category, no label).
  Participants
    Infants: <=18 years | 73 | 0 | 73
    Infants: Between 18 and 65 years | 0 | 73 | 73
    Infants: >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 14 | 48
  Male | 39 | 59 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 10 | 23
  Not Hispanic or Latino | 59 | 63 | 122
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 59 | 64 | 123
  More than one race | 8 | 3 | 11
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Infant Visual Attention
Description: Infant visual attention was measured for all 3 conditions using head mounted eye-tracking. Duration of visual attention (total duration of infant visual fixations greater than 100 ms each, to the book during shared book reading) was measured within a spatial window of the scene. Proportations of visual attention to the book were calculated by dividing attention duration to the book by the total task duration
Time Frame: Day 1
Population: One infant was excluded due to equipment failure, 9 infants excluded due to unwillingness to wear the eye-tracking equipment, and 2 excluded for test dates falling outside the 28 day age group exclusion window.
Measure: Mean (Standard Deviation); unit: Proportion of Visual Attention Duration
Groups:
- Effects of Shared Book Reading: Effect of Labels 6 Month Olds: Proportions of visual attention to the book were calculated by dividing attention duration to the book by the total task duration for the 6 month olds.
- Effects of Shared Book Reading: Labels 9 Month Olds: Proportions of visual attention to the book were calculated by dividing attention duration to the book by the total task duration for the 9 month olds.
- Effects of Shared Book Reading: Labeling 12 Month Olds: Proportions of visual attention to the book were calculated by dividing attention duration to the book by the total task duration for the 12 month olds.
Arm/Group | Effects of Shared Book Reading: Effect of Labels 6 Month Olds | Effects of Shared Book Reading: Labels 9 Month Olds | Effects of Shared Book Reading: Labeling 12 Month Olds
Number analyzed (Participants) | 20 | 21 | 18
Proportion of Visual Attention Duration
  Individual | .533 (.206) | .358 (.157) | .377 (.252)
  Category | .544 (.236) | .300 (.168) | .351 (.226)
  No Label | .472 (.222) | .257 (.174) | .404 (.207)
Statistical Analysis 1: Comparison: Effects of Shared Book Reading: Effect of Labels 6 Month Olds vs Effects of Shared Book Reading: Labels 9 Month Olds vs Effects of Shared Book Reading: Labeling 12 Month Olds; To examine the impact of infant age and label condition on the proportion of infant's attention to the book, a 3 (infant age: 6, 9, or 12 months) x 3 (label condition: individual, categorical, or no label) MANOVA was run. Age was measured between subjects, label condition was within subjects, and infant's proportion of attention to the book was the dependent variable. The main effect of age is reported here; Test type: Superiority; p = .002, MANOVA — F(2, 58) = 7.19
Statistical Analysis 2: Comparison: Effects of Shared Book Reading: Effect of Labels 6 Month Olds vs Effects of Shared Book Reading: Labels 9 Month Olds vs Effects of Shared Book Reading: Labeling 12 Month Olds; To examine the impact of infant age and label condition on the proportion of infant's attention to the book, a 3 (infant age: 6, 9, or 12 months) x 3 (label condition: individual, categorical, or no label) MANOVA was run. Age was measured between subjects, label condition was within subjects, and infant's proportion of attention to the book was the dependent variable. The main effect of condition is reported here; Test type: Superiority; p = .09, MANOVA — F(1.78, 103.37) = 2.48
Statistical Analysis 3: Comparison: Effects of Shared Book Reading: Effect of Labels 6 Month Olds vs Effects of Shared Book Reading: Labels 9 Month Olds vs Effects of Shared Book Reading: Labeling 12 Month Olds; To examine the impact of infant age and label condition on the proportion of infant's attention to the book, a 3 (infant age: 6, 9, or 12 months) x 3 (label condition: individual, categorical, or no label) MANOVA was run. Age was measured between subjects, label condition was within subjects, and infant's proportion of attention to the book was the dependent variable. The interaction between age and condition is reported here; Test type: Superiority; p < .05, MANOVA — F(3.56, 103.37) = 2.55

2. Primary Outcome: Infant EEG Steady-state Evoked Potential Frequency Tagging Power
Description: To examine the extent to which infant EEG power, as measured by the signal-to-noise ratio (SNR) was modulated by label condition and age, data were extracted from a mid-occipital cluster of Oz and its 6 nearest neighbors (channels 70, 71, 74, 75, 76, 82, 83) for each of the conditions by age group.
Time Frame: On Day 2
Population: Two dyads were excluded for technical issues during EEG recording, and 5 dyads who completed visit one but did not have EEG data collected.
Measure: Mean (Standard Deviation); unit: Signal to Noise Ratio
Groups:
- Effects of Shared Book Reading: Labeling 6 Month Olds: 6-month old infant EEG power for objects from all three conditions.
- Effects of Shared Book Reading: Labeling 9 Month Olds: 9-month old infant EEG power for objects from all three conditions.
- Effects of Shared Book Reading: Labeling 12 Months: 12-month old infant EEG power for objects from all three conditions.
Arm/Group | Effects of Shared Book Reading: Labeling 6 Month Olds | Effects of Shared Book Reading: Labeling 9 Month Olds | Effects of Shared Book Reading: Labeling 12 Months
Number analyzed (Participants) | 15 | 17 | 19
Signal to Noise Ratio
  Individual | 7.270 (.856) | 7.506 (.642) | 7.392 (.639)
  Category | 7.298 (.606) | 7.583 (.670) | 7.108 (.603)
  No Label | 7.256 (.879) | 7.449 (.728) | 7.612 (.570)
Statistical Analysis 1: Comparison: Effects of Shared Book Reading: Labeling 6 Month Olds vs Effects of Shared Book Reading: Labeling 9 Month Olds vs Effects of Shared Book Reading: Labeling 12 Months; EEG power, as measured by the signal-to-noise ratio (SNR) was modulated by label condition across age, data were extracted from a mid-occipital cluster of Oz and its 6 nearest neighbors (channels 70, 71, 74, 75, 76, 82, 83) for each of the conditions. SNR data were then submitted to a two-factor MANOVA with Label (Individual, Category, Control/No Label) as a within-subjects factor and Age (6 months, 9 months, 12 months) as a between-subjects factor. The main effect of age is reported here; Test type: Superiority; p = .557, MANOVA — F(2,47) = .592
Statistical Analysis 2: Comparison: Effects of Shared Book Reading: Labeling 6 Month Olds vs Effects of Shared Book Reading: Labeling 9 Month Olds vs Effects of Shared Book Reading: Labeling 12 Months; EEG power, as measured by the signal-to-noise ratio (SNR) was modulated by label condition across age, data were extracted from a mid-occipital cluster of Oz and its 6 nearest neighbors (channels 70, 71, 74, 75, 76, 82, 83) for each of the conditions. SNR data were then submitted to a two-factor MANOVA with Label (Individual, Category, Control/No Label) as a within-subjects factor and Age (6 months, 9 months, 12 months) as a between-subjects factor. The main effect of condition is reported here; Test type: Superiority; p = .470, MANOVA — F(2,47) = .767
Statistical Analysis 3: Comparison: Effects of Shared Book Reading: Labeling 6 Month Olds vs Effects of Shared Book Reading: Labeling 9 Month Olds vs Effects of Shared Book Reading: Labeling 12 Months; EEG power, as measured by signal-to-noise ratio (SNR) was modulated by label condition across age, data were extracted from a mid-occipital cluster of Oz and its 6 nearest neighbors (channels 70, 71, 74, 75, 76, 82, 83) for each condition. SNR data were then submitted to a two-factor MANOVA with Label (Individual, Category, Control/No Label) as a within-subjects factor and Age (6 months, 9 months, 12 months) as a between-subjects factor. The interaction of age and condition is reported here; Test type: Superiority; p = .046, MANOVA — F(4,94) = 2.524

3. Secondary Outcome: Infant and Parent EEG Synchrony
Description: Infant and parent EEG synchrony (as a dyad) was quantified and compared across conditions. We used a phase-locking index to quantify EEG dyadic synchrony across conditions. The phase-locking index measures the extent to which the parent and infant oscillatory response is in the same phase across time. This index is bounded between 0 and 1, with 1 being perfect synchrony.
Time Frame: On Day 2
Population: The data represent the number of dyads (infant plus 1 parent) analyzed. Dyads were excluded for technical issues during EEG recording and 5 dyads were excluded because they completed visit 1 but did not have EEG data collected for Visit 2.
Measure: Mean (Standard Deviation); unit: Phase Locking Index
Groups:
- Effects of Shared Book Reading: Labeling 6 Month Olds: Infant (6-month-old) and parent EEG synchrony (as a dyad) was quantified and compared across conditions.
- Effects of Shared Book Reading: Labeling 9 Month Olds; Effects of Shared Book Reading: Labeling 12 Months: Infant (9-month-old) and parent EEG synchrony (as a dyad) was quantified and compared across conditions.
Arm/Group | Effects of Shared Book Reading: Labeling 6 Month Olds | Effects of Shared Book Reading: Labeling 9 Month Olds | Effects of Shared Book Reading: Labeling 12 Months
Number analyzed (Participants) | 15 | 17 | 19
Phase Locking Index
  Individual Label | .478 (.053) | .484 (.048) | .461 (.037)
  Categorical Label | .471 (.048) | .488 (.043) | .474 (.034)
  No Label | .471 (.063) | .480 (.043) | .480 (.034)
Statistical Analysis 1: Comparison: Effects of Shared Book Reading: Labeling 6 Month Olds vs Effects of Shared Book Reading: Labeling 9 Month Olds vs Effects of Shared Book Reading: Labeling 12 Months; EEG Data were extracted from a mid-occipital cluster for each conditions for parents & infants. Data were entered into a 2-factor MANOVA with Label (Individual, Category, No Label) as a within-subjects factor and Age (6 mo, 9 mo, 12 mo) as a between-subjects factor. The phase-locking index measures the extent to which the parent & infant oscillatory response is in the same phase across time (bounded between 0 and 1, 1 being perfect synchrony. The main effect of age is reported here; Test type: Superiority; p = .664, MANOVA — F(2,45) = .413
Statistical Analysis 2: Comparison: Effects of Shared Book Reading: Labeling 6 Month Olds vs Effects of Shared Book Reading: Labeling 9 Month Olds vs Effects of Shared Book Reading: Labeling 12 Months; EEG Data were extracted from a mid-occipital cluster for each conditions for parents & infants. Data were entered into a 2-factor MANOVA with Label (Individual, Category, No Label) as a within-subjects factor and Age (6 mo, 9 mo, 12 mo) as a between-subjects factor. The phase-locking index measures the extent to which the parent & infant oscillatory response is in the same phase across time (bounded between 0 and 1, 1 being perfect synchrony. The main effect of condition is reported here; Test type: Superiority; p = .768, MANOVA — F(2,45) = .266
Statistical Analysis 3: Comparison: Effects of Shared Book Reading: Labeling 6 Month Olds vs Effects of Shared Book Reading: Labeling 9 Month Olds vs Effects of Shared Book Reading: Labeling 12 Months; EEG Data were extracted from a mid-occipital cluster for each conditions for parents & infants. Data were entered into a 2-factor MANOVA with Label (Individual, Category, No Label) as a within-subjects factor and Age (6 mo, 9 mo, 12 mo) as a between-subjects factor. The phase-locking index measures the extent to which the parent & infant oscillatory response is in the same phase across time (bounded between 0 and 1, 1 being perfect synchrony. The interaction of age and condition is reported; Test type: Superiority; p = .200, MANOVA — F(4,90) = 1.531

4. Secondary Outcome: Parent-Infant Visual Joint Attention
Description: Parent and infant visual attention (as a dyad) was measured across conditions using dual parent and infant head mounted eye-tracking. Duration of joint attention (periods of overlap of parent and infant visual fixations to the book during shared book reading) was measured within a spatial window of the scene. Proportions of joint attention were calculated by dividing joint attention duration by the total task duration.
Time Frame: On Day 1
Population: The data represent the number of dyads analyzed. 60 dyads (27 Female Infants, 33 Male Infants; 47 Female caregivers; 13 Male Caregivers) were included in the final sample. The final sample included dyads with 20 6-month infants, 23 9-month infants, and 17 12-month infants.
Measure: Mean (Standard Deviation); unit: Joint Attention Proportion Mean
Groups:
- Effects of Shared Book Reading: Labeling 6 Month Olds; Effects of Shared Book Reading: Labeling 9 Month Olds: 6-month old infants and a parent completed shared book reading and proportion of joint visual attention (dyad, co-occurrence of parent and infant attention toward the book) was measured across conditions.
- Effects of Shared Book Reading: Labeling 12 Month Olds: 12-month old infants and a parent completed shared book reading and proportion of joint visual attention (dyad, co-occurrence of parent and infant attention toward the book) was measured across conditions.
Arm/Group | Effects of Shared Book Reading: Labeling 6 Month Olds | Effects of Shared Book Reading: Labeling 9 Month Olds | Effects of Shared Book Reading: Labeling 12 Month Olds
Number analyzed (Participants) | 20 | 23 | 17
Joint Attention Proportion Mean
  Individual | .356 (.170) | .262 (.145) | .286 (.219)
  Category | .409 (.210) | .222 (.150) | .276 (.198)
  No Label | .323 (.176) | .180 (.167) | .254 (.179)
Statistical Analysis 1: Comparison: Effects of Shared Book Reading: Labeling 6 Month Olds vs Effects of Shared Book Reading: Labeling 9 Month Olds vs Effects of Shared Book Reading: Labeling 12 Month Olds; To examine the impact of infant age and label condition on the proportion of joint attention to the book, a 3 (infant age: 6, 9, or 12 months) x 3 (label condition: individual, categorical, or no label) MANOVA was run. Age was measured between subjects, label condition was within subjects, and the proportion of joint attention to the book was the dependent variable. The main effect of age is reported here; Test type: Superiority; p = .022, MANOVA — F(2, 57) = 4.11
Statistical Analysis 2: Comparison: Effects of Shared Book Reading: Labeling 6 Month Olds vs Effects of Shared Book Reading: Labeling 9 Month Olds vs Effects of Shared Book Reading: Labeling 12 Month Olds; To examine the impact of infant age and label condition on the proportion of joint attention to the book, a 3 (infant age: 6, 9, or 12 months) x 3 (label condition: individual, categorical, or no label) MANOVA was run. Age was measured between subjects, label condition was within subjects, and the proportion of joint attention to the book was the dependent variable. The main effect of condition is reported here; Test type: Superiority; p = .004, MANOVA — F(2, 114) = 5.69
Statistical Analysis 3: Comparison: Effects of Shared Book Reading: Labeling 6 Month Olds vs Effects of Shared Book Reading: Labeling 9 Month Olds vs Effects of Shared Book Reading: Labeling 12 Month Olds; To examine the impact of infant age and label condition on the proportion of joint attention to the book, a 3 (infant age: 6, 9, or 12 months) x 3 (label condition: individual, categorical, or no label) MANOVA was run. Age was measured between subjects, label condition was within subjects, and the proportion of joint attention to the book was the dependent variable. The interaction of age and condition is reported here; Test type: Superiority; p = .168, MANOVA — F(4, 114) = 1.64

ADVERSE EVENTS:
Time Frame: Solicited adverse events were collected through day 2, unsolicited adverse events were collected up to 6 months
Description: Defined by NIH criteria.
Groups:
- Effects of Shared Book Reading: There will be one arm since all participants will undergo the same intervention.
  Book reading: Parent and their infant will read a short book in the laboratory. Books will include three labeling conditions expected to elicit different levels of attention.
Arm/Group | Effects of Shared Book Reading
All-Cause Mortality (participants affected / at risk) | 0/146
Serious Adverse Events (participants affected / at risk) | 0/146
Other Adverse Events (participants affected / at risk) | 0/146

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT04337372/Prot_001.pdf
  • Informed Consent Form (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT04337372/ICF_000.pdf